CLINICAL TRIAL: NCT00882141
Title: Menopause, Genes and Metabolism After Weight Loss and Exercise
Brief Title: Race, Menopause and Metabolism After Exercise and Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Alice S. Ryan, Ph.D., University of Maryland School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0116; R01AG019310 (NIH); R01AG020116 (NIH)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Insulin Resistance; Sedentary Lifestyle
Keywords: Exercise; Obesity; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance; Sedentary Behavior; Motor Activity | interventions — Diet Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Weight loss
  Interventions: Behavioral: Diet modification
- 2 (Experimental): Exercise plus weight loss
  Interventions: Behavioral: Diet modification; Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Diet modification — Weight loss sessions are held by a registered dietitian for 1 hour once a week for 6-9 months; recommended caloric intake to elicit a weight loss of approximately 0.2-0.4 kg per week
  Other Names: American Heart Association "Heart Healthy" diet
Behavioral: Aerobic exercise — Treadmills and other aerobic exercise equipment 3 times a week for 6-9 months, beginning at low levels of VO2max and progressing in duration and intensity to more than 75% VO2max for 45 minutes
  Arms: 2

SUMMARY:
The purpose of this study is to test the hypotheses that there are ethnic and genetic differences in the mechanisms and magnitude by which hypocaloric weight loss and aerobic exercise affect body composition, glucose, lipid, muscle and adipose tissue metabolism in overweight, insulin resistant postmenopausal women. This will be tested in a trial comparing the effects of weight loss vs. aerobic exercise plus weight loss on glucose, lipid, fat and muscle metabolism in overweight African American and Caucasian postmenopausal women.

DETAILED DESCRIPTION:
The findings of this study will also determine whether there are racial differences in the whole body and cellular mechanisms by which aerobic exercise training and weight loss affect glucose, lipid, fat and muscle metabolism in African-American vs. Caucasian postmenopausal women. The results also may provide a rationale for targeting specific populations of women who might improve glucose, lipid, fat and muscle metabolism more from the addition of exercise to dietary restriction than weight loss alone to reduce their risk for type 2 diabetes and cardiovascular disease.

The study protocol consists of the following phases:

Phase 1-Recruitment and screening.

Phase 2-Weight and dietary stabilization for 4-6 weeks, where participants are taught the principles of the American Heart Association "Heart Healthy" diet and provided food to consume prior to testing.

Phase 3-Participants will undergo research testing including glucose clamp and fat biopsy.

Phase 4-Participants select either weight loss only, or exercise plus weight loss. The behavior diet modification weight loss sessions are held by a registered dietitian for 1 hour once a week for 6-9 months where the recommended caloric intake for each participant is adjusted by the dietitian to elicit a weight loss of approximately 0.2-0.4 kg per week. In addition to the weight loss sessions, participants who select the aerobic exercise plus weight loss intervention will exercise at the Baltimore Geriatric Research Education and Clinical Center (GRECC) exercise facility 3 times a week for 6-9 months using treadmills and other aerobic exercise equipment. Exercise sessions begin at low levels of VO2max (maximal oxygen consumption) and progress in duration and intensity until the participant is able to exercise at more than 75% VO2max for 45 minutes.

Phase 5-Following the 6-9 months of long-term weight loss or exercise plus weight loss, all participants will undergo long-term metabolic testing.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45-80 yrs of age
* Non-smoking for one year
* BMI greater than 25 kg/m2 and less than 50 kg/m2
* Menopause over 1 year
* Caucasian or African American ethnicity

Exclusion Criteria:

Both groups

* Currently being treated for active cancer
* Type 1 diabetes; insulin treatment; poorly controlled (fasting blood sugar over 160 mg/dl)
* Allergic to lidocaine or heparin
* Untreated dyslipidemia, receiving triglyceride-lowering meds
* Other systemic disorders that are not medically treated and stable
* Taking beta-blockers, oral steroids, warfarin or any other medications interfering with fat/muscle metabolism that may not be safely discontinued temporarily for specific procedures (i.e. for 72 hours prior)
* Abnormal liver or renal function; chronic pulmonary disease (on supplemental oxygen); anemia
* MMSE (Mini-Mental State Examination) below 24, dementia or unstable clinical depression by exam
* Women of ethnicity other than Caucasian or African American
* Symptomatic heart disease, coronary artery disease, congestive heart failure, or uncontrolled hypertension unless medically stabilized
* Abnormal response to exercise test (chest pain, significant arrhythmias, extreme shortness of breath, cyanosis, exercising blood pressure above 240/120mm Hg, or other contraindications to exercise)

Exercise plus weight loss group only

* Medical history of CVD (cardiovascular disease) with symptoms limiting ability to exercise
* Physical impairment limiting normal activity
* Aerobically trained with VO2max greater than 2 SD (standard deviation) above age-adjusted mean

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2002-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Glucose Clamp | At 4-6 weeks
Fat biopsy | At 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — University of Maryland, VA Research Service; Andrew P. Goldberg, MD, Principal Investigator — University of Maryland, VA Research Service
Locations (1):
- University of Maryland, VAMC, Baltimore, Maryland, United States

REFERENCES:
- [Background] Berman DM, Rodrigues LM, Nicklas BJ, Ryan AS, Dennis KE, Goldberg AP. Racial disparities in metabolism, central obesity, and sex hormone-binding globulin in postmenopausal women. J Clin Endocrinol Metab. 2001 Jan;86(1):97-103. doi: 10.1210/jcem.86.1.7147. PMID 11231984
- [Background] Ryan AS, Nicklas BJ, Berman DM. Racial differences in insulin resistance and mid-thigh fat deposition in postmenopausal women. Obes Res. 2002 May;10(5):336-44. doi: 10.1038/oby.2002.47. PMID 12006632
- [Background] Nicklas BJ, Dennis KE, Berman DM, Sorkin J, Ryan AS, Goldberg AP. Lifestyle intervention of hypocaloric dieting and walking reduces abdominal obesity and improves coronary heart disease risk factors in obese, postmenopausal, African-American and Caucasian women. J Gerontol A Biol Sci Med Sci. 2003 Feb;58(2):181-9. doi: 10.1093/gerona/58.2.m181. PMID 12586858
- [Background] Ryan AS, Nicklas BJ, Berman DM. Aerobic exercise is necessary to improve glucose utilization with moderate weight loss in women. Obesity (Silver Spring). 2006 Jun;14(6):1064-72. doi: 10.1038/oby.2006.122. PMID 16861612
- [Derived] Ryan AS, Serra MC, Goldberg AP. Metabolic Benefits of Prior Weight Loss with and without Exercise on Subsequent 6-Month Weight Regain. Obesity (Silver Spring). 2018 Jan;26(1):37-44. doi: 10.1002/oby.22032. Epub 2017 Oct 25. PMID 29071802
- [Derived] Ortmeyer HK, Goldberg AP, Ryan AS. Exercise with weight loss improves adipose tissue and skeletal muscle markers of fatty acid metabolism in postmenopausal women. Obesity (Silver Spring). 2017 Jul;25(7):1246-1253. doi: 10.1002/oby.21877. Epub 2017 May 26. PMID 28547918
- [Derived] Ge S, Ryan AS. Zinc-alpha2-glycoprotein expression in adipose tissue of obese postmenopausal women before and after weight loss and exercise + weight loss. Metabolism. 2014 Aug;63(8):995-9. doi: 10.1016/j.metabol.2014.04.013. Epub 2014 May 4. PMID 24929893
- [Derived] Ryan AS, Ge S, Blumenthal JB, Serra MC, Prior SJ, Goldberg AP. Aerobic exercise and weight loss reduce vascular markers of inflammation and improve insulin sensitivity in obese women. J Am Geriatr Soc. 2014 Apr;62(4):607-14. doi: 10.1111/jgs.12749. Epub 2014 Mar 17. PMID 24635342
- [Derived] Prior SJ, Blumenthal JB, Katzel LI, Goldberg AP, Ryan AS. Increased skeletal muscle capillarization after aerobic exercise training and weight loss improves insulin sensitivity in adults with IGT. Diabetes Care. 2014 May;37(5):1469-75. doi: 10.2337/dc13-2358. Epub 2014 Mar 4. PMID 24595633
- [Derived] Yang RZ, Blumenthal JB, Glynn NM, Lee MJ, Goldberg AP, Gong DW, Ryan AS. Decrease of circulating SAA is correlated with reduction of abdominal SAA secretion during weight loss. Obesity (Silver Spring). 2014 Apr;22(4):1085-90. doi: 10.1002/oby.20657. Epub 2013 Dec 6. PMID 24311467
- [Derived] Ryan AS, Li G, Blumenthal JB, Ortmeyer HK. Aerobic exercise + weight loss decreases skeletal muscle myostatin expression and improves insulin sensitivity in older adults. Obesity (Silver Spring). 2013 Jul;21(7):1350-6. doi: 10.1002/oby.20216. Epub 2013 May 19. PMID 23687104